CLINICAL TRIAL: NCT06067165
Title: Primary Care Online Emotion-regulation Treatment (POET)
Acronym: POET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Region Skane (Other); Region Östergötland (Other); Västra Götalandsregionen (Other)
Responsible Party: Principal Investigator, Johan Bjureberg, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-03652-01
Record Dates: First submitted 2023-09-17; First posted 2023-10-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mental Health Issue
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting post- and follow-up assessments will be blind to treatment allocation, for the full duration of the trial. The outcome measures are identical for both groups, ensuring that the assessors remain blind. To ensure blinding integrity, participants receive explicit instructions not to disclose which treatment participants have received. After completing the assessment, the blind raters guess the participant's group allocation and disclose the reason for their guess and record whether the participants has inadvertently revealed their group allocation. Blind assessments will be recorded to allow for calculation of inter-rater reliability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POET feeling (Experimental): POET will include six guided digital treatment modules for the youth, and six modules for the parents administered over the course of six weeks.
  Interventions: Behavioral: POET feeling
- Supportive treatment (Active Comparator): The active control will be supportive treatment. It includes six guided digital treatment modules for the youth, and six modules for the parents administered over the course of six weeks.
  Interventions: Behavioral: Supportive treatment

INTERVENTIONS:
Behavioral: POET feeling — POET is adapted from online Emotion Regulation Individual Therapy for Adolescents developed by the research group (ClinicalTrials.gov Identifier: NCT03353961).
  POET is also based on the Modal model of emotion and Process model of emotion regulation that provides a framework for understanding how emotions are generated, experienced and how they can be regulated. The youth component of POET will include psychoeducation, addressing maladaptive beliefs about emotions and emotion regulation, and teaching adaptive emotion regulation strategies, such as acceptance of emotions and flexible cognitive reappraisal. The parent component will include psychoeducation and teaching effective support and responding to their adolescent's and their own emotions.
  Arms: POET feeling
Behavioral: Supportive treatment — The treatment will include educative material on mental health and self-reflection on themes such as school, family and friends. The parent component will include educative material and self reflection in how to support their adolescent.
  Arms: Supportive treatment

SUMMARY:
Mental health problems in youth are a global problem, causing incalculable suffering in youth and families, harming long-term prospects of youths, and creating substantial economic costs to society.

The overall objective of this study is to build an evidence base for a highly scalable transdiagnostic intervention called the Primary care Online Emotion-regulation Treatment (POET) for youth (12-17 years) seeking treatment for mental health problems.

In a randomized controlled trial, the investigators will examine the effects of POET. The investigators will test if emotion regulation mediates reduction in mental health problems during treatment. In addition the investigators will test if POET is more effective for some individuals than others and evaluate if POET is cost-effective. The investigators will also test whether there are detectable effects of POET on distal outcomes utilizing registry data following participants up to 10 years post treatment.

DETAILED DESCRIPTION:
Introduction:

Mental health problems among young people are prevalent and many youth in need of treatment for mental health problems do not meet criteria for any mental health disorder or they meet criteria for several disorders. Most existing treatments focus on a subset of mental disorders and do not address subthreshold or multi-disorder mental health problems. In addition, available treatments do not typically target transdiagnostic disease mechanisms. Furthermore, the available treatments are limited in efficacy and most youth in need do not receive treatment due to social stigma and structural barriers such as geographical distance to treatment providers.

The aim of this randomized clinical trial is to determine the clinical efficacy of a digital emotion regulation treatment in adolescents with mental health problems. Participants will be randomized to a digital emotion regulation treatment or to an active comparator. Treatments in both conditions will include therapist support, and will be delivered in a blended treatment format combining asynchronous therapist-guided online modules with one synchronous session delivered over video-link. The primary endpoint is at post- treatment.

Primary objectives:

1. To test the effects of POET on mental health problems.
2. To test the effects of POET on emotion regulation.

Secondary objectives:

1. To test if emotion regulation mediates reductions in mental health problems during treatment.
2. To test if POET is cost-effective.
3. To test if POET works better for some individuals than others (i.e., moderation).
4. To test if there are detectable differences in distal outcomes between POET and active control 12 to 60 months post treatment and if individual baseline characteristics moderates these effects.

Research questions:

1. What are the effects of POET on mental health problems?
2. What are the effects of POET on emotion regulation?
3. Are reductions in mental health problems during the POET treatment mediated through emotion regulation?
4. Is POET feeling cost-effective?
5. Does POET work better for some individuals than others?
6. Are there detectable differences in distal outcomes between POET and active control 12 to 60 months post treatment and if individual baseline characteristics moderates these effects

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 - 17 years
* Seeking care for mental health problems
* At least one guardian interested in participating in the parent program
* Deemed capable of making decisions

Exclusion Criteria:

* Psychiatric problems that require more extensive treatment.
* Low global functioning (under 41 points on clinician rated C-GAS or functioning that requires more extensive treatment).
* Elevated suicide risk
* Insufficient Swedish comprehension.
* Life circumstances that complicate or make treatment impossible (eg severe deficits in parental care, domestic violence).
* Change in psychopharmacological medication in the last 2 months.
* Ongoing psychological treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 388 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2031-11-25 (Estimated)

PRIMARY OUTCOMES:
The Clinical Global Impressions -Severity scale (CGI-S) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess symptom severity rated on a single item ranging from 1-7, with higher scores indicating more severe symptoms. Clinician-rated.

SECONDARY OUTCOMES:
The Clinical Global Impressions - Improvement scales (CGI-I) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess symptom improvement rated on a single item ranging from 1-7, with lower scores indicating more improvement. Clinician-rated.
The Revised Child Anxiety and Depression Scale-C (RCADS-C) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess symptoms of depression and anxiety. This scale has 47 items, total score ranging from 0 to 141, with higher scores indicating more severe symptoms. Clinician-rated.
The Revised Child Anxiety and Depression Scale-P (RCADS-P) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess symptoms of depression and anxiety in their offspring. This scale has 47 items, total score ranges from 0 to 141 points, with higher scores indicating more severe symptoms. Caregiver-reported.
Brief 11-item version of the Revised Child Anxiety and Depression Scale for Adolescents (RCADS-11) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess symptoms of depression and anxiety in children and adolescents. This scale has 11 items, total score ranges from 0-33 points, with higher scores indicating more severe symptoms. Self-rated by adolescents.
Children's global assessment scale (CGAS) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess global impairment on a single item ranging from 1 to 100, with a higher value indicating better functioning. Clinician-rated.
The Work and Social Adjustment Scale (WSAS) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess impaired functioning in school, everyday life, friends and social life, recreation and hobbies and family and close relationships. This scale has 5 items, total score ranges from 0 to 40, with higher scores indicating greater impairment. Clinician-rated.
The Positive and Negative Affect Schedule for Children (PANAS-C) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess positive and negative feelings. This scale has 2 subscales. Each total subscale score range from 5-25, with higher scores indicating more negative or positive feelings. Self-rated by adolescents.
The Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess cognitive reappraisal. The subscale has 6 items, total subscale score ranges from 6-30, with higher scores indicating greater usage of cognitive reappraisal. Self-rated by adolescents.
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess difficulties in emotion regulation. The scale has 16 items, total score ranges from 16-80, with higher scores indicating more difficulties. Self-rated by adolescents.
  One subscale named impulse (3 items ranging from 3-15) will be administered once every week during treatment.
The Process Model of Emotion Regulation Questionnaire -short (PMERQ-S) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assesses individual differences in emotion regulation. This scale has 30 items, total score ranges from 30-180, with higher scores indicate a greater usage of emotion regulation. Self-rated by adolescents.
  The three subscales named Confront unpleasant situations (3 items, total subscale score ranges from 6-18), Avoid unpleasant situations (3 items, total subscale score ranges from 6-18) and Cognitively distract (3 items, total subscale score ranges 6-18) will administered to adolescents weekly.
The Perth Alexithymia Questionnaire-Short Form (PAQ-S) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess alexithymia. This scale has 6 items, total score ranges from 6 to 42, with higher scores indicate higher levels of alexithymia. Self-rated by adolescents.
Self-Efficacy Questionnaire for Children (SEQ-C) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7 after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess social self-efficacy. The subscale named social self-efficacy has 8 items, total subscale score ranges from 8-40, with higher scores indicating greater social self-efficacy. Self-rated by adolescents.
Child Health Utility 9D (CHU-9D) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess health-related quality of life. This scale has 9 items, total score ranges from 9 to 45, with higher scores indicating worse quality of life. Self-rated by adolescents.
Borderline symptoms checklist supplement (BSL-23) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess high-risk and problematic behaviors. This scale has 10 items, total score ranges from 0 to 40, with higher scores indicating greater usage of high-risk and problematic behaviors. Self-rated by adolescents.
The Emotion Beliefs Questionnaire (EBQ) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess beliefs about emotions. This scale 16 items, total score ranges from 16 to 112, with higher scores indicating more maladaptive beliefs about emotions. Self-rated by adolescents.
Coping with Children's Negative Emotions Scale Adolescent Version (CCNES-A) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess parents' perceived ability to cope with children's negative emotions. This scale has six subscales which include emotion focused, problem-focused, minimization, punitive, expressive encouragement, and distress responses. Each subscale has 9 items, total subscale score ranges from 1-7, with higher scores indicating greater usage of a certain parental coping style. Care-giver reported.
Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess difficulties in emotion regulation. The scale has 16 items, total score ranges from 16-80, with higher scores indicating more difficulties. Self-rated by parents.
Behavioral emotion regulation questionnaire (BERQ) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess parents' perception of the adolescent's behavioral emotion regulation. This scale has 5 subscales. Each total subscale score ranges from 4-20, with higher scores indicating greater usage of a certain strategy. Care-giver reported.
Trimbos Questionnaire for Costs associated with Psychiatric Illness (TiC-P) | Week 0, 7 weeks after treatment start and 3,12 and 60 months after treatment has ended
  Used to assess healthcare and other societal resource use for both children and caregivers. Caregiver-reported.
Deliberate Self-Harm Inventory, Youth version (DSHI-Y) | 3,12 and 60 months after treatment has ended
  Used to assess occurrence, method, frequency of deliberate self-harm. This scale has 6 items with higher scores indicating more frequent deliberate self-harm. Self-rated by adolescents.

OTHER OUTCOMES:
The Credibility/Expectancy Questionnaire (CEQ) | Week 0 and Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 after treatment start.
  Used to assess treatment credibility and expectancy. The scale has 5 items ranging from 4-58 with higher scores indicating greater credibility/expectancy. Clinician-reported, adolescents self-rated, care-giver reported.
Client Satisfaction Questionnaire (CSQ) | 7 weeks after treatment start
  Used to assess client satisfaction with treatment. This scale has 8 items ranging from 8-32 points with higher scores indicating greater treatment satisfaction. Adolescents self-rated, care-giver reported.
Patient Internet Cognitive behavior therapy Adherence Scale (PIAS) | 3 and 7 weeks after treatment start
  Used to assess patient adherence to internet-delivered behavioral interventions. This scale has 5 items, total score ranging from 0 to 20, where 0 indicates no adherence and 20 perfect adherence. Clinician-rated.
Questionnaire on Adverse events | 7 weeks after treatment start
  Used to assess adverse events related to treatment. Adolescents are asked to report any negative effects or adverse events throughout the treatment period. Adolescents are also requested to report the extent of the impact of any potential adverse events on their well-being using a 0-4 scale, with a higher score indicating a more significant impact. Adolescent self-reported.
Academic performance | 5 years after after treatment has ended
  Grades in school using data from the Swedish registry Longitudinal Integration Database for Health Insurance and Labour Market Studies (LISA).
Occupation | 5 years after after treatment has ended
  Unemployment rates using data from the Swedish registry Longitudinal Integration Database for Health Insurance and Labour Market Studies (LISA) that contains information on occupation.
Health-care consumption | 5 years after after treatment has ended
  Number of health care visits using data from the National (Sweden) Patient Register.
Psychopharmacological treatment | 5 years after after treatment has ended
  Number of psychotropic medications using data from National (Sweden) Prescribed Drug Register.
Mental health disorders | 5 years after after treatment has ended
  Number of mental disorders according to the ICD-10 and ICD-11 using data from the National (Sweden) Patient Register.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Bjureberg, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The data are pseudonymized according to national (Swedish) and European Union legislation and cannot be anonymized and published in an open repository. Participants in the study consent for their data to be shared with other international researchers for meta-analyses. Aggregated data can be made available upon reasonable request on a case-by-case basis according to the current legislation and ethical permits